CLINICAL TRIAL: NCT00089752
Title: Impact of CPAP on Functional Outcomes in Milder Obstructive Sleep Apnea (CATNAP)
Brief Title: Continuous Positive Airway Pressure to Improve Milder Obstructive Sleep Apnea
Acronym: CATNAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Respironics Sleep and Respiratory Foundation (Unknown); Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 163; R01HL076101 (NIH)
Record Dates: First submitted 2004-08-12; First posted 2004-08-16 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Lung Diseases; Sleep Apnea Syndromes; Hypertension
MeSH Terms: conditions — Lung Diseases; Sleep Apnea Syndromes; Hypertension | interventions — Continuous Positive Airway Pressure; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Treatment (Active Comparator): Continuous Positive Airway Pressure Treatment
  Interventions: Device: Continuous Positive Airway Pressure (CPAP) Treatment
- Sham/Placebo Treatment (Placebo Comparator): Ineffective sham continuous positive airway pressure device with leak in interface to <1.0 cm H2O and resistance in motor to simulate normal operating noise and no compensation for leak.
  Interventions: Device: Sham CPAP device - CPAP device with pressure delivered <1 cm H20

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) Treatment — CPAP device used at night
  Other Names: Positive Airway Pressure
  Arms: Active Treatment
Device: Sham CPAP device - CPAP device with pressure delivered <1 cm H20 — Sham CPAP device used at night
  Arms: Sham/Placebo Treatment

SUMMARY:
The purpose of this study is to determine whether functional status improves in individuals with milder obstructive sleep apnea (OSA) following continuous positive airway pressure (CPAP) treatment.

DETAILED DESCRIPTION:
BACKGROUND:

OSA is characterized as mild, moderate, or severe, according to the number of respiratory disturbances per hour of sleep (RDI), as defined by the American Academy of Sleep Medicine. CPAP is the primary treatment for sleep apnea. The column of pressure delivered to the upper airway by this device immediately eliminates the respiratory disturbances when it is applied. There is evidence from randomized controlled studies that CPAP also improves functional status, and the key manifestation of OSA, including excessive daytime sleepiness, in individuals with severe OSI (i.e., RDI greater than 30). However, there has been limited research exploring improvement in functional status in individuals with less severe OSA (i.e., those with mild OSA and RDI of 5-15 or moderate OSA and RDI of 16-30). The large placebo effect that has been reported in controlled studies of OSA-associated functional outcomes mandates the need for a placebo in studies evaluating the true impact of this treatment. Results from the three randomized controlled studies in milder OSA that have examined this issue have been equivocal, principally because of serious methodological limitations. It remains unclear whether CPAP treatment improves daily functioning in those with milder OSA (RDI 5-30). This is a critical issue as this level of disease severity represents the largest segment of OSA and comprises 15% of the U.S. population.

DESIGN NARRATIVE:

Using Granger's model of functional assessment, this study will examine whether functional status improves in participants with milder OSA following CPAP treatment. The study will employ a randomized, placebo-controlled, parallel study design, and will use a sham CPAP device as the placebo in participants with significant daytime sleepiness. The study will test the hypothesis that the change in functional status (measured by the Functional Outcomes of Sleep Questionnaire) after 8 weeks of treatment will be greater for participants treated with active CPAP compared to the placebo. Secondary aims of the study include examining whether CPAP also improves daytime sleepiness, and determining whether CPAP can reduce nocturnal blood pressure to lower the risk for stroke and hypertension linked to OSA.

ELIGIBILITY:
Inclusion Criteria

* Newly diagnosed with OSA on overnight polysomnogram (PSG) with RDI between 5 and 30
* Score of greater than 11 on the Epworth Sleepiness Scale (ESS) on two administrations of the instrument (performed at prescreening and screening), each completed on a different day to avoid sporadic values and confirm the presence of excessive daytime sleepiness
* Stable medical history and no change in medications, including hypertension medications, in the 3 months prior to study entry
* Stable psychiatric history and no change in psychotropic medications in the 3 months prior to study entry
* Has access to a telephone

Exclusion Criteria

* Diagnosis of another sleep disorder in addition to OSA based on PSG, e.g., periodic limb movement disorder (greater than 10 limb movements per hour of sleep with arousal); central sleep apnea (greater than 5 or more central apneas); insomnia; sleep hypoventilation syndrome; or narcolepsy
* Previous treatment for sleep apnea with nasal CPAP, oral appliance, home oxygen therapy, uvulopalatopharyngoplasty, tracheotomy, or other surgery for OSA
* Oxygen or bi-level CPAP required for treatment of OSA
* Unable to return for study instructions or follow-up testing
* Medically unstable condition (e.g., heart attack, congestive heart failure, Cheyne-Stokes breathing, unstable angina, uncontrolled thyroid disease, unstable diabetes, depression or psychosis, ventricular arrhythmias, cirrhosis, or recently diagnosed cancer) in the 3 months prior to study entry
* Regular use (greater than 3 times per week) of sedative, hypnotic, or alerting medications (such as Modafinil) in the 3 months prior to study entry
* Chronic nasal congestion that would prevent the use of a nasal mask, in the 3 months prior to study entry
* History of automobile accidents due to excessive daytime sleepiness
* Employed in transportation-related safety sensitive occupation such as an airline pilot, truck driver, or train engineer
* Night shift worker regularly experiencing jet lag, or a history of irregular work schedules in the 6 months prior to study entry
* Regular use of alcohol as determined by answering yes to one or more of the questions on the CAGE questionnaire (i.e., alcohol dependent)
* Recent or recurring history of substance abuse leading to tolerance or dependence
* Pregnant; women must either be postmenopausal or confirmed not pregnant by a urine pregnancy test
* Unable to perform study tests, e.g., inability to communicate verbally; inability to write and read in English; less than a 5th grade reading level (evaluated using Flesch-Kincaid assessment); visual impairment; hearing impairment; cognitive impairment (e.g., previous head injury); or upper extremity motor deficit (e.g., previous stroke or spinal cord injury)
* Residing with an individual who is currently using CPAP treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2003-09; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri Weaver, Study Chair — University of Pennsylvania
Locations (5):
- United States (4):
  - National Jewish Medical and Research Center (NJC), Denver, Colorado
  - Emory University School of Medicine (EMO), Atlanta, Georgia
  - North Shore-Long Island Jewish Health System (LIJ), Long Island City, New York
  - New York University Medical School, New York, New York
- University of Western Ontario (UWO), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Petition of Principal Investigator with document outlining purpose of secondary analysis and use of the data, which is then reviewed with co-investigators for overall approval.

REFERENCES:
- [Result] Weaver TE, Mancini C, Maislin G, Cater J, Staley B, Landis JR, Ferguson KA, George CF, Schulman DA, Greenberg H, Rapoport DM, Walsleben JA, Lee-Chiong T, Gurubhagavatula I, Kuna ST. Continuous positive airway pressure treatment of sleepy patients with milder obstructive sleep apnea: results of the CPAP Apnea Trial North American Program (CATNAP) randomized clinical trial. Am J Respir Crit Care Med. 2012 Oct 1;186(7):677-83. doi: 10.1164/rccm.201202-0200OC. Epub 2012 Jul 26. PMID 22837377
- [Derived] Rodway GW, Weaver TE, Mancini C, Cater J, Maislin G, Staley B, Ferguson KA, George CF, Schulman DA, Greenberg H, Rapoport DM, Walsleben JA, Lee-Chiong T, Kuna ST. Evaluation of sham-CPAP as a placebo in CPAP intervention studies. Sleep. 2010 Feb;33(2):260-6. doi: 10.1093/sleep/33.2.260. PMID 20175410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the sleep disorders clinic from each of the 5 participating centers. Potential participants were approached by study staff at each site once their medical record indicated that they may be candidates for the study. Recruitment commenced 1-11-05 and ended 4-18-2008.
Groups:
- Active CPAP: Continuous positive pressure device that delivers therapeutic positive airway pressure to maintain airway patency worn continuously for each night of treatment.
- Sham CPAP: A device that looks and sounds like an active continuous positive pressure device (CPAP) that delivers ineffective pressure, i.e.,less than 1 cm H20 pressure compared to greater than 5 cm H20 for active treatment. Like active CPAP treatment it is worn every night.
Period: Overall Study
Arm/Group | Active CPAP | Sham CPAP
Started | 141 | 140
Completed | 121 | 118
Not Completed | 20 | 22

BASELINE CHARACTERISTICS:
Groups:
- Active CPAP: CPAP device
- Sham CPAP: Sham CPAP device
- Total: Total of all reporting groups
Arm/Group | Active CPAP | Sham CPAP | Total
Number analyzed (Participants) | 121 | 118 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 116 | 112 | 228
  >=65 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 44 | 99
  Male | 66 | 74 | 140
Region of Enrollment [Number; unit: participants]
  United States | 68 | 68 | 136
  Canada | 53 | 50 | 103

OUTCOME MEASURES:

1. Primary Outcome: Change in the Score of the Functional Outcomes of Sleep Questionnaire at Baseline and Week 8 Treatment
Description: The primary endpoint is change after 8 weeks of treatment from baseline value (controlling for baseline value) in the 30-item Functional Outcomes of Sleep Questionnaire (FOSQ) that will be used to test the primary study hypothesis that patients with milder OSA (RDI 5-30) on active treatment will demonstrate greater mean change for the Total score from baseline to 8 weeks treatment. The FOSQ is designed to assess the impact of excessive sleepiness on functional status. The instrument has established content validity, test-retest reliability (r= 0.91), and internal consistency (alpha = 0.96). The scale ranges from 5 - 20 with normal functional status being a value greater than 17.
Time Frame: 8 weeks
Population: Consented and randomized participants who completed the FOSQ with mild or moderate obstructive sleep apnea.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Active CPAP: continuous positive airway pressure device
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 121 | 118
scores on a scale | 0.98 (2.89) | -0.14 (2.61)

2. Secondary Outcome: Change in the Score From Baseline to 8 Weeks Treatment Epworth Sleepiness Scale
Description: Change in the score from baseline to 8 weeks treatment, controlling for baseline in the self-rated 8 item measure of daytime sleepiness with a range from 0 - 24. Lower values indicting less daytime sleepiness
Time Frame: Measured at Baseline and Week 8 of treatment in ITT sample
Population: Participants randomized and who had post-treatment data in ITT analysis
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- CPAP: Active Continuous Positive Airway Pressure device
- Shame CPAP: Ineffective (placebo) Continuous Positive Airway Pressure device
Arm/Group | CPAP | Shame CPAP
Number analyzed (Participants) | 105 | 102
scores on a scale | -2.58 (4.28) | -0.54 (3.49)

3. Secondary Outcome: Change in Mean Arterial Daytime Pressure at Baseline and Week 8 Treatment
Description: Change in mean arterial pressure (MAP) value from baseline to 8 weeks treatment, controlling for baseline, measured by 48 hours ambulatory blood pressure device - Space Laboratories
Time Frame: Measured at Baseline and Week 8 treatment in the ITT sample
Population: Population who had data post-randomization following 8 wks. intervention - ITT analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CPAP | Shame CPAP
Number analyzed (Participants) | 80 | 72
mmHg | 90.3 (7.6) | 92 (7.9)
Statistical Analysis 1: Comparison: CPAP vs Shame CPAP; Intent to Treat analysis with Last Observation Carried Forward; Test type: Non-Inferiority or Equivalence — Sample size was designed to achieve at least 80% power, using n 1⁄4 123 per group with an effect size of at least 0.36; p = 0.09, ANCOVA — a priori threshold was p<0.05; Adjusted difference in mean change = -1.76, 95% CI 2-sided [-3.8 to 0.3]

4. Secondary Outcome: Change in the Score From Baseline to 8 Weeks Treatment Measured by the Profile of Mood States
Description: Change in the score from baseline to 8 weeks treatment, controlling for baseline, in the POMS is a reliable and valid measure of mood states that consists of 65 adjectives on which subjects' rate themselves as they feel "today" using a five-point scale. There are six mood or affective states on this test derived through factor analysis: Tension-Anxiety (score range 0-36), Depression-Dejection (score range 0 - 60), Anger-Hostility (score range 0-48), Vigor-Activity (score range 0-32), Fatigue-Inertia (score range 0-28), and Confusion-Bewilderment (score range 0-28). There is also a summary Total Mood Disturbance (TMD) score that gives a Total estimate of affective state score range 0-200). Higher scores indicate greater disability.
Time Frame: Measured at Baseline and Week 8 treatment in the ITT sample
Population: Population who had data post-randomization following 8 wks. intervention - ITT analysis
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CPAP | Shame CPAP
Number analyzed (Participants) | 107 | 103
scores on a scale | -10.2 (25.5) | -0.5 (20.1)

5. Secondary Outcome: Change in the Number of Lapses From Baseline to 8 Weeks Treatment on the Psychomotor Vigilance Task (PVT) - Total Lapses in 20 Minute Test
Description: Change in the score from baseline to 8 weeks treatment, controlling for baseline, in the PVT is an objective assessment of sleepiness and measures decrements in neurobehavioral performance due to sleepiness, i.e., ability to sustain attention and respond in a timely manner to salient signals.(7) The PVT yields five highly informative metrics on the capacity for sustained attention and vigilance performance: frequency of lapses, duration of lapse domain, optimum response time, vigilance decrement function, false response frequency. We applied this conceptually valid, relatively short duration, reliable task with known psychometric properties and minimal practice/learning curves to document attentional lapses (response times > 500 msec) in performance.
Time Frame: Baseline and 8 weeks of treatment in the ITT sample
Population: The Intent-to-Treat Sample includes all randomized patients receiving at least a 20 minute interval of Active during the post randomization treatment period and who had no clinically significant major violations of inclusion or exclusion criteria.
Measure: Mean (Standard Deviation); unit: number on a scale
Arm/Group | CPAP | Shame CPAP
Number analyzed (Participants) | 102 | 96
number on a scale | -2.91 (26.12) | 2.99 (21.54)

6. Secondary Outcome: Change in the Score From Baseline to 8 Weeks Treatment on the SF36 - Physical
Description: Change in the score from baseline to 8 weeks treatment, controlling for baseline, in the SF-36 is a 36-item questionnaire that assesses eight health concepts: physical functioning, bodily pain, role limitations due to physical problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Higher scores indicate greater disability with a range of scores from 0-100.
Time Frame: Baseline and Week 8 of treatment in ITT sample.
Population: The Intent-to-Treat Sample includes all randomized patients exposed to CPAP or Sham treatment during the post randomization treatment period.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CPAP | Shame CPAP
Number analyzed (Participants) | 84 | 85
scores on a scale | 3.92 (7.46) | -0.19 (6.99)

7. Secondary Outcome: Change in the Score From Baseline to 8 Weeks Treatment SF-36 Mental Component
Description: as for outcome 6
Time Frame: Baseline and after 8 weeks of treatment in ITT sample
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CPAP | Shame CPAP
Number analyzed (Participants) | 84 | 85
scores on a scale | 3.38 (9.83) | 2.00 (8.10)

ADVERSE EVENTS:
Time Frame: 5 years
Description: From beginning of recruitment until study termination (5 years) . All non-serious adverse events reported and unspecified relative to whether it was associated with the intervention.
Groups:
- Active CPAP: Continuous positive pressure device that delivers therapeutic (prescribed > 5 CM H2O) positive airway pressure worn continuously for each night of treatment for 8 wks.
- Sham CPAP: A device worn continuously every night that looks and sounds like an active continuous positive pressure device (CPAP) that delivers ineffective pressure, i.e.,less than 1 cm H20 pressure for 8 wks.
Arm/Group | Active CPAP | Sham CPAP
Serious Adverse Events (participants affected / at risk) | 6/121 | 11/118
Other Adverse Events (participants affected / at risk) | 93/121 | 94/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active CPAP (N=121) | Sham CPAP (N=118)
Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 3 (4) — TOOTH DISORDER VOMITING No relation to study
Cardiac (Cardiac disorders) | 1 (1) | 2 (2) — Arrhythmia, palpitations General cardiac Chest pain No relation to study
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — SOFT TISSUE FRACTURE No relation to study
Pain (Nervous system disorders) | 1 (1) | 0 (0) — HEADACHE - No relation to study
Constitutional Symptoms (General disorders) | 1 (1) | 0 (0) — Pyrexia - No relation to study
Renal (Renal and urinary disorders) | 0 (0) | 1 (1) — Prostatic obstruction - No relation to study
Dermatology/Skin (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) — No relation to study
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — UPPER RESPIRATORY-Possibly related to study
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (2) — Upper GI Epistaxis - possibly related to study
Blood/Bone Marrow (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Low hemoglobin - No relation to study
Infection (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Clostridial infection - No relation to study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active CPAP (N=121) | Sham CPAP (N=118)
Rhinitis Allergic nos/ Allergy Other-Possibly related to study (Immune system disorders) | 27 (28) | 35 (35) — MedDRA codes provided in the CTC AE (Publish date: December 12, 2003) correspond with MedDRA 6.0
Dermatology/Skin - Possibly related to study (Skin and subcutaneous tissue disorders) | 20 (20) | 22 (22) — Mask irritation of the skin Dermatitis exfoliative nos Dermatology/skin - other Ecchymosis
Constitutional Symptoms (General disorders) | 4 (25) | 9 (9) — Fatigue - Possibly related to study Insomnia
Gastrointestinal (Gastrointestinal disorders) | 15 (23) | 21 (36) — Abdominal distention- Possibly related to study Constipation Diarrhea nos Dry mouth- Possibly related to study Dyspepsia Gastrointestinal - other Nausea - Possibly related to study Vomiting nos
Infection - Not related to study (Infections and infestations) | 14 (24) | 25 (47) — Sinus infection Upper aerodigestive Upper airway Not study related
Musculoskeletal/Soft Tissue- Not related to study (Musculoskeletal and connective tissue disorders) | 7 (8) | 10 (15) — Upper extremity/function Soft tissue
Neurology - Not related to study (Nervous system disorders) | 7 (9) | 10 (12) — Anxiety Dizziness Neurology-other
Pain- possibly related to study (General disorders) | 47 (102) | 51 (116) — Arthralgia, back pain, chest wall pain, facial pain,headache, neck pain, oral pain, pain - other, pain in extremity, pharyngolary pain, sinus pain, stomach discomfort, toothache
Pulmonary/Upper Respiratory - Possibly related to study (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 15 (22) — Bronchospasm Cough, Nasal cavity/paranasal sinus pulmonary/upper respiratory
Syndromes - Not related to study (Infections and infestations) | 1 (1) | 8 (12) — Influenza-like illness

LIMITATIONS AND CAVEATS:
Post-randomization adverse events are summarized by treatment arm & body system.The CTC-AE (Publish Date December 12, 2003) was utilized for coding verbatim (raw) adverse event data with a MedDRA code, Body System, AE/Supraordinate term & Grade.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No